CLINICAL TRIAL: NCT00300924
Title: A Double-Blind, Double-Dummy, Randomized, Parallel-Group, Placebo Controlled Study to Evaluate the Efficacy and Tolerability of Rizatriptan 10mg Co-Administered With Acetaminophen for the Treatment of Acute Migraine.
Brief Title: A Study of Rizatriptan Co-Administered With Acetaminophen for the Treatment of Acute Migraine
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Diamond Headache Clinic (Other)
Collaborators: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Karin E. Brooks, BSN, RN Director of Clinical Research, Diamond Headache Clinic
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: Merck 075-00; Merk 075-00
Record Dates: First submitted 2006-03-09; First posted 2006-03-10 (Estimated); Last update posted 2008-05-28 (Estimated); Status verified 2008-05

CONDITIONS: Migraine
MeSH Terms: conditions — Migraine Disorders | interventions — Acetaminophen

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Drug: Rizatriptan co-administered with Acetaminophen

SUMMARY:
The purpose of this study is to test an experimental drug combination of two medications currently approved by the Food and Drug Administration (FDA) for migraine headache or other pain. These are called rizatriptan given with acetaminophen.

ELIGIBILITY:
Inclusion Criteria:

* Subject is at least 18 years of age
* Subject has at least a 6 month history of migraine, with or without aura
* Subject can distinguish between migraine attacks and other types of headaches
* Subject of childbearing potential agrees to use adequate contraception

Exclusion Criteria:

* Subject typically has fewer than 1 or greater than 6 migraine attacks per month
* Subject typically has greater than 10 headache days per month
* Subject has evidence of ischemic heart disease
* Subject has uncontrolled high blood pressure
* Subject has a history, within 1 year, or current evidence of drug or alcohol abuse

*This list is not all inclusive*

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200
Dates: Start 2006-03; Primary Completion 2007-01 (Actual); Study Completion 2007-01 (Actual)

PRIMARY OUTCOMES:
To compare the efficacy of rizatriptan co-administered with acetaminophen to placebo, acetaminophen and rizatriptan for the acute treatment of migraine, as measured by the percentage of patients with pain relief at 2 hours.

SECONDARY OUTCOMES:
24 hour sustained pain relief
Pain relief at 30, 45,60,90 minutes and 4 hours post dose
Pain freedom at 30,45,60,90 minutes and 2 and 4 hours post dose
24 sustained pain freedom
Associated symptoms of phonophobia, photophobia, nausea and vomiting
Functional disability
Use of rescue medication
Self-reported adverse experiences

CONTACTS AND LOCATIONS:
Overall Officials: Merle Diamond, M.D., Study Director — Diamond Headache Clinic
Locations (7):
- United States (7):
  - SanFrancisco Headache Clinic, San Francisco, California
  - Diamond Headache Clinic, Chicago, Illinois
  - Westside Family Medical Center, Kalamazoo, Michigan
  - Clinvest, Springfield, Missouri
  - Mercy Health Research, St Louis, Missouri
  - Elkind Headache Center, Mount Vernon, New York
  - ClinExcel, West Chester, Ohio